CLINICAL TRIAL: NCT00490399
Title: A Phase II Trial of GEMZAR Combined With Cisplatin in Patients With Inoperable Biliary Tract Carcinomas
Brief Title: Trial of Gemcitabine and Cisplatin in Patients With Inoperable Biliary Tract Carcinomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6689; B9E-KL-S292
Record Dates: First submitted 2007-06-20; First posted 2007-06-22 (Estimated); Last update posted 2007-06-22 (Estimated); Status verified 2007-06

CONDITIONS: Biliary Tract Carcinoma
MeSH Terms: interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: gemcitabine
Drug: cisplatin

SUMMARY:
The purpose of this study is to evaluate the efficacy of gemcitabine and cisplatin in Korean patients with biliary tract (bile tracts of the gallbladder or liver) cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of adenocarcinoma of the gallbladder, intra/extrahepatic bile ducts or papilla of Vater with locally advanced or metastatic disease (at study entry) that is not amenable to curative surgical resection or with recurrent disease after prior surgical resection or radiotherapy.
* Disease status must be measurable disease defined as: Bi-dimensionally measurable lesions with clearly defined margins and two perpendicular diameters that are clearly measurable by following:

  * Computerized tomography (CT) or magnetic resonance imaging (MRI), with one diameter 2.0 cm or greater and the other diameter 1.0 cm or greater.
  * Palpable Lesion, with both diameters 2 cm or greater. Disease progressing in areas of prior radiation therapy may be included.
* Patients must have received no prior chemotherapy for advanced disease.
* Prior radiotherapy must be completed at least 4 weeks before study enrollment. Patients must have recovered from the acute toxic effects of the treatment prior to study enrollment.

Exclusion Criteria:

* Treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Heart failure, angina pectoris or arrhythmia that are poorly controlled in spite of medication or acute myocardial infarction within 6 months preceding study enrollment
* Severe neurological or mental disorder.
* Active infection that in the opinion of the investigator would compromise the patient's ability to tolerate therapy.
* Poorly controlled diabetes mellitus.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2003-03; Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the response rate

SECONDARY OUTCOMES:
To characterize the quantitative and qualitative toxicities of gemcitabine combined with cisplatin in this patient population.
To evaluate the following time-to-event efficacy variables: Duration of response, Time to treatment failure, Time to documented disease progression, Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul, South Korea

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com